CLINICAL TRIAL: NCT02049476
Title: Proof of Concept Study of the Effectiveness of Ozurdex in Lieu of Oral Corticosteroids for the Control of Active Intermediate and Posterior Uveitis Requiring Immunosuppressive Drug Therapy
Brief Title: Study of the Effectiveness of Ozurdex for the Control of Uveitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00088146
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Uveitis, Intermediate; Uveitis, Posterior
Keywords: Uveitis, Intermediate; Uveitis, Posterior; Dexamethasone; Immunosuppressive Agents; Eye Abnormalities; Eye Diseases; Ophthalmology; Ophthalmologic Surgical Procedures; Vision Disorders; Inflammation
MeSH Terms: conditions — Uveitis, Intermediate; Uveitis, Posterior; Eye Abnormalities; Eye Diseases; Vision Disorders; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone Pellet (Experimental): This is a proof of concept study; therefore all enrolled patients will receive the intervention according to its FDA-approved indication.
  Interventions: Drug: Dexamethasone pellet

INTERVENTIONS:
Drug: Dexamethasone pellet — Dexamethasone pellet placement occurs within 14 days of baseline examination; for patients with bilaterally active uveitis, placement of a dexamethasone pellet in the second eye should occur within 14 days of the first implantation or within 30 day of the baseline examination.
  Repeated placement is permitted every 3 months based on the best clinical judgment of the doctor and the study protocol.
  Other Names: Ozurdex pellet

SUMMARY:
The main purpose of this study is to evaluate whether or not the dexamethasone pellet (Ozurdex®, Allergan, Irvine, CA) can replace oral corticosteroid (e.g. prednisone) in the treatment of active sight-threatening, noninfectious intermediate and/or posterior uveitis in which immunosuppressive drug therapy is indicated.

Uveitis is an inflammation inside the eye. Uveitis can decrease patients' vision if it is not treated.

The dexamethasone pellet is an implant filled with a corticosteroid medicine. This therapy is approved by the Food and Drug Administration (FDA) for the treatment of intermediate and/or posterior uveitis.

In this study investigators want to see if using the implant together with systemic immunosuppressive drug therapy can result in lower ocular side effect profile but is effective enough to replace the use of high-dose systemic corticosteroids in the treatment of active intermediate and/or posterior uveitis. Knowing the effectiveness and safety of these treatments is important because the kinds of uveitis being studied usually need to be treated for many years. This information may help researchers understand uveitis better and may suggest ways of improving treatment.

Adult patients with intermediate and/or posterior uveitis for which immunosuppressive drug therapy with high-dose corticosteroid is planned may join.

DETAILED DESCRIPTION:
Objectives: This is a single arm study evaluating whether or not the dexamethasone pellet (Ozurdex®, Allergan, Irvine, CA) can replace oral corticosteroid (e.g. prednisone) in the treatment of active sight-threatening, noninfectious intermediate or posterior uveitis in which immunosuppressive drug therapy is indicated.

Background: Intermediate and posterior uveitis are thought to be severe intraocular inflammation that may lead to permanent visual loss. It is estimated that these forms of uveitis comprise the fifth or sixth leading cause of blindness and tend to affect working class age patients, thus causing loss of work hours and diminished productivity and quality of life. Because the posterior segment of the eye is not adequately treated by corticosteroid drops often systemic drug therapy is used including oral corticosteroids or prednisone. Prednisone can have a myriad of side effects in approximately one-quarter to one-third of cases treated in tertiary care centers such as ours, additional medications such as immunosuppressive drugs are required to control the disease and/or to allow for appropriate tapering of oral prednisone to subsequent levels that have a low side effect profile when delivered over a long period of time. Typically, chronic prednisone therapy in doses of 7.5 mg daily or less are thought to have a low enough side effect profile to be amenable to long-term therapy. However frequently immunosuppressive drugs are required to get the dosing to this level. There are occasions when patients are intolerant of any dose of oral corticosteroids or are intolerant of the higher doses of oral corticosteroids (30 - 60 mg daily) and therefore this treatment modality is avoided due to prednisone's attendant side effects. Although periocular and intravitreal corticosteroids injections may be performed, with these modalities the standard of care is to wait until the disease reactivates before instituting such therapy and therefore a chronic suppressive dose is not obtained. The fluocinolone acetonide implant (Retisert®, Bausch and Lomb, Tampa, FL) is FDA-approved for the treatment of intermediate and posterior uveitis and it is equally effective in controlling uveitis as high-dose oral corticosteroids but avoids the systemic side effects associated with the use of high doses of oral corticosteroids. However, this form of local therapy has high rates of ocular side effects, including ocular hypertension causing glaucoma and/or requiring glaucoma surgery and cataracts. Furthermore, every two and half to three years the implant is exhausted of corticosteroid and therefore repeat surgical insertion of another implant may be required. A useful potential therapy for the treatment of these patients would be a shorter-acting local corticosteroid that could be delivered in conjunction with systemic immunosuppressive drug therapy that would have a lower ocular side effect profile but still would be effective enough to replace the use of high-dose systemic corticosteroids in the treatment of active intermediate or posterior uveitis. It is possible that the dexamethasone pellet could fill this unique role in the treatment of uveitis. Investigators propose this study to evaluate dexamethasone pellet for this specific use among patients with active intermediate and posterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Active sight-threatening intermediate or posterior uveitis for which immunosuppressive drug therapy is planned and the physician is considering treatment with high-dose corticosteroid to control the uveitis whilst immunosuppressive drugs are being instituted or adjusted. Note: it is acceptable for the patient to already be on an immunosuppressive drug as long as high dose corticosteroids are indicated.
* Patients must be age 18 years or older (the dexamethasone pellet is not FDA-approved for pediatric use) and sign an informed consent.
* The ocular media must be clear enough to obtain optical coherence photography (OCT) and fundus photographs.
* No elective intraocular surgery should be planned for the first 3 months after enrollment.

Exclusion Criteria:

* Infectious uveitis
* History of scleritis
* Active or suspected viral infection of the cornea or conjunctiva
* History of mycobacterial or fungal disease
* HIV positivity
* Age <18 years old
* Allergy to dexamethasone
* Uncontrolled intraocular pressure (IOP)
* Advanced glaucoma
* Aphakia with rupture of the posterior lens capsule
* Anterior chamber IntraOcualr Lens (ACIOL) with rupture of the posterior lens capsule
* Media opacity that would preclude evaluation of the posterior pole via fundus photography or OCT assessment
* Planned elective ocular surgery within 3 months of enrollment
* Any systemic disease requiring systemic corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Thorne, MD, PhD, Principal Investigator — Department of Ophthalmology, Johns Hopkins School of Medicine,
Locations (1):
- The Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Dexamethasone Pellet: This is a proof of concept study; therefore all enrolled patients will receive the intervention according to its FDA-approved indication.
  Dexamethasone pellet: Dexamethasone pellet placement occurs within 14 days of baseline examination; for patients with bilaterally active uveitis, placement of a dexamethasone pellet in the second eye should occur within 14 days of the first implantation or within 30 day of the baseline examination.
  Repeated placement is permitted every 3 months based on the best clinical judgment of the doctor and the study protocol.
Period: Overall Study
Arm/Group | Dexamethasone Pellet
Started | 20; 28 Eyes (First patient enrolled on 1/31/2014)
Completed | 20; 28 Eyes (20th patient completed the study)
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Dexamethasone Pellet
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Type of uveitis [Count of Participants; unit: Participants] — Type of uveitis is determined by the primary anatomic location of the inflammation.
  Participants
    Anterior and Intermediate | 7
    Intermediate | 4
    Posterior | 9
Bilaterality of uveitis [Count of Participants; unit: Participants] — Defined as either unilateral (one eye) or bilateral (both eye) with active uveitis.
  Participants
    Unilateral | 0
    Bilateral | 20
Activity of uveitis [Count of Participants; unit: Participants] — Active disease as defined by treating ophthalmologist. Typically this is active vitreous cell or vitreous haze in the case of intermediate uveitis and active chorioretinal lesions or retinal vasculitis/leakage in posterior uveitis.
  Participants
    Active vitreous cell | 8
    Active vitreous haze | 4
    Active chorioretinal lesions | 2
    Active retinal vasculitis/leakage | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Intraocular Inflammation at 6 Months
Description: Absence of intraocular inflammation (e.g. less than trace anterior chamber (AC) cells; no vitreous haze; inactive chorioretinal lesions) is used to assess control of intraocular inflammation following treatment.
Time Frame: at 6-month visit
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Pellet
Number analyzed (Participants) | 20
Participants | 12

2. Secondary Outcome: Number of Participants With Absence of Intraocular Inflammation at 12 Months
Description: as for outcome 1
Time Frame: 12-month clinical visit
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Pellet
Number analyzed (Participants) | 20
Participants | 13

3. Other Pre Specified Outcome: Mean Intraocular Pressure (IOP)
Description: Mean IOP (mmHg) was calculated at each visit
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months visit
Measure: Mean (Standard Deviation); unit: millimeters of Mercury (mm Hg)
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Pellet
Number analyzed (Participants) | 20
Number analyzed (eyes) | 28
millimeters of Mercury (mm Hg)
  Baseline IOP | 13.2 (0.8)
  Month 1 Visit | 18.2 (2.0)
  Month 3 Visit | 14.6 (1.3)
  Month 6 Visit | 14.1 (1.3)
  Month 12 Visit | 13.5 (1.1)

4. Other Pre Specified Outcome: Number of Eyes With a Need for Cataract Surgery
Description: Number of eyes that had progression of cataract defined as any interval increase in nuclear, cortical or posterior sub capsular cataract from a previous visit that resulted in cataract surgery.
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months visit
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Pellet
Number analyzed (Participants) | 20
Number analyzed (eyes) | 28
eyes
  Baseline visit | 0
  Month 1 visit | 0
  Month 3 visit | 0
  Month 6 visit | 1
  Month12 visit | 3

ADVERSE EVENTS:
Time Frame: All 20 patients were followed for 12 months after their first Ozurdex injection to look for adverse events
Arm/Group | Dexamethasone Pellet
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Pellet (N=20)
Cataract progression (Eye disorders) | 4 (6)
Ocular hypertension (Eye disorders) | 7 (9) — Intraocular pressure (IOP) of 25 mmHg or higher on any visit
Cataract surgery (Eye disorders) | 2 (4) — progression of a cataract that required surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02049476/Prot_SAP_000.pdf